CLINICAL TRIAL: NCT07397832
Title: CRP Regimen (Chidamide, Rituximab and Polatuzumab Vedotin) in Treating Elderly Patients With Previously Untreated Double-Positive DLBCL: Single-Arm, Open-Label, Multicenter Phase II Trial
Brief Title: CRP Regimen in Treating Elderly Patients With Previously Untreated Double-Positive DLBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Huilai Zhang, Study director, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRP-DLBCL01
Record Dates: First submitted 2026-01-04; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Diffuse Large B-Cell Lymphoma (DLBCL)
Keywords: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Rituximab; polatuzumab vedotin; pola office

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination therapy with Chidamide, Rituximab and Polatuzumab VedotinCRP Regimen + Chidamide Mainten (Experimental): Each subject will be given combination therapy of Chidamide, Rituximab and Polatuzumab Vedotin.The maximum number of treatment cycles is six.
  Interventions: Drug: Chidamide; Drug: Rituximab; Drug: Polatuzumab Vedotin; Drug: Chidamide Maintenance

INTERVENTIONS:
Drug: Chidamide — Chidamide: patients followed a step-dose escalation regimen (10mg BIW,15mg BIW, 20mg BIW). 21 days as a treatment cycle. The maximum number of treatment cycles is six.
  Other Names: HDACi
Drug: Rituximab — Day 1 of each cycle, 375 mg/m².The maximum number of treatment cycles is six.
  Other Names: R
Drug: Polatuzumab Vedotin — Day 1 of each cycle, 1.8 mg/kg. The maximum number of treatment cycles is six.
  Other Names: Pola
Drug: Chidamide Maintenance — For patients assessed as being in PR or CR status after completion of combination therapy, maintenance therapy with chidamide is administered for one year at a dosage of 20 mg, BIW. Drug adjustments may be made based on the patient's tolerance, with reference to the drug prescribing information.
  Other Names: HDACi Maintenance

SUMMARY:
A Single-Arm, Open-Label, Multicenter Phase II Trial of CRP Regimen (Chidamide, Rituximab, Polatuzumab Vedotin) in Treating Elderly Patients with Previously Untreated Double-Positive Diffuse Large B-Cell Lymphoma

DETAILED DESCRIPTION:
This is a single-arm, open-label, multicenter Phase II trial to evaluate the feasibility, efficacy, and safety of the CRP regimen (Chidamide, Rituximab, Polatuzumab Vedotin) in treating elderly patients with previously untreated double-expressor diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥70 years, or patients aged 60-69 years with an ECOG performance status score of 2-4. Both males and females are eligible.
2. No prior treatment for DLBCL, including chemotherapy, targeted therapy, immunotherapy, local radiotherapy directed at the lymphoma (excluding palliative radiotherapy for symptom relief), or surgical therapy (excluding diagnostic biopsy or surgery not targeting the lymphoma).
3. Histopathological confirmation meeting all of the following conditions:

   1. Diagnosis of diffuse large B-cell lymphoma (DLBCL) with CD20 positivity; concurrent positive expression of C-MYC and Bcl-2 (double-expressor phenotype).
   2. At least one measurable lesion positive on ¹⁸F-FDG PET-CT scan according to the Lugano 2014 criteria for Hodgkin and non-Hodgkin lymphoma.
4. Laboratory tests at screening must meet the following criteria, unless the investigator attributes abnormalities to lymphoma (no corrective or supportive therapy for these parameters within 2 weeks prior to assessment):

   1. Hematology: Hb ≥90 g/L, ANC ≥1.5 × 10⁹/L, PLT ≥90 × 10⁹/L.
   2. Biochemistry: Cr ≤1.5 ×ULN; TBIL ≤1.5 × ULN; ALT and AST ≤2.5 × ULN (for patients with liver involvement: ≤5 × ULN).
5. Life expectancy of at least 6 months, as judged by the investigator.
6. Ability to understand and voluntarily provide written informed consent.

Exclusion Criteria:

1. History of or concurrent other active malignancies.
2. Prior treatment with Chidamide and/or R-CHOP. Contraindication to any component of CHOP, including prior anthracycline therapy. History of severe hypersensitivity or anaphylaxis to humanized or murine monoclonal antibodies, or known sensitivity/allergy to murine products.
3. Current diagnosis of any of the following: Follicular lymphoma grade 3B; B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and classical Hodgkin lymphoma (grey zone lymphoma); Primary mediastinal (thymic) large B-cell lymphoma; Burkitt lymphoma; Central nervous system (CNS) lymphoma (primary or secondary); Primary effusion DLBCL; Primary cutaneous DLBCL, leg type.
4. History of myocardial infarction, unstable angina, or other clinically significant cardiac disease within 12 months prior to signing informed consent; or prior coronary angioplasty/stenting within 12 months.
5. Clinically uncontrolled active infection (bacterial, fungal, or viral) or organ hemorrhage.
6. Pregnant or lactating women.
7. Participation in any other clinical trial within 6 months prior to signing informed consent.
8. Any other condition that, in the opinion of the investigator, makes the patient unsuitable for participation in this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CRR) | up to the end of CRP Regimen treatment, no more than 6 cycles, each cycle is 21 days
  To assess the Complete Response Rate (CR) at the end of CRP Regimen (Chidamide, Rituximab, Polatuzumab Vedotin).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | up to the end of CRP Regimen treatment, no more than 6 cycles, each cycle is 21 days
  To assess the Overall Response Rate (ORR) at the end of CRP Regimen (Chidamide, Rituximab, Polatuzumab Vedotin).
Progression-free survival (PFS) | up to 2 years
  The time from study enrollment to the first documented disease progression or death from any cause, whichever occurs first."
Event free survival(EFS) | up to 2 years
  The duration from the time of study enrollment until the occurrence of disease progression, relapse after complete response (CR), death from any cause, or the initiation of new treatment for residual lesions after completion of combination therapy (including switched therapy for lesions during the trial), whichever occurs first.
Overall Survival(OS) | up to 2 years
  The time from subject enrollment to Death caused by any reason. for patients lost to follow-up, the time of the last follow-up; for patients still alive at the end of study, the date of the end of follow-up.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.The frequency and severity of adverse events were evaluated based on changes in various vital sign indicators and laboratory tests.
Quality of Life Assessment - EORTC QLQ-C30 Score | up to 2 years
  Quality of life will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). The score changes in overall quality of life, functional scales, and symptom scales will be analyzed in relation to clinical outcomes.
Quality of Life Assessment - FACT-Lym Score | up to 2 years
  Disease-specific quality of life will be assessed using the Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) questionnaire (Version 4). The score changes will be analyzed in relation to clinical outcomes.

OTHER OUTCOMES:
Biomarkers Associated with Treatment Response and Disease Progression | up to 2 years
  Using Whole Transcriptome Sequencing (WTS) and Next-Generation Sequencing (NGS), we will examine if baseline molecular/proteomic subtypes, genomic profiles, and specific somatic mutations affect CRP regimen efficacy or drive disease progression to more severe states.
Biomarkers Associated with Adverse Events | up to 2 years
  We will use Whole Transcriptome Sequencing (WTS) and NGS to investigate whether specific somatic mutations increase the risk of CRP regimen-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Huilai Zhang, Study Director — Tianjin Medical University Cancer Insititute & Hospital
Locations (1):
- Tianjin Medical University Cancer Insititute & Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No